CLINICAL TRIAL: NCT03104439
Title: Nivolumab and Ipilimumab and Radiation Therapy in Microsatellite Stable (MSS) and Microsatellite Instability (MSI) High Colorectal and Pancreatic Cancer
Brief Title: Nivolumab and Ipilimumab and Radiation Therapy in MSS and MSI High Colorectal and Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Julie Koenig, Physician, Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-021
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Microsatellite Stable Colorectal Cancer; Pancreatic Cancer; MSI High Colorectal Cancer
Keywords: Pancreatic Cancer; Microsatellite Stable Colorectal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Ipilimumab (Experimental): * Nivolumab will be administered intravenously 3 times per cycle
  * Ipilimumab will be administered intravenously once per cycle
  * Radiation Therapy will be administered per hospital standard
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — The antibodies in nivolumab work by causing programmed cell death of the cancer cells
  Other Names: Opdivo
Drug: Ipilimumab — The antibodies in ipilimumab work by not allowing cancer cell growth
  Other Names: Yervoy
Radiation: Radiation Therapy — Radiation therapy is believed to increase the likelihood of response of immunotherapy

SUMMARY:
This research study is studying a combination of drugs with radiation therapy as a possible treatment for Microsatellite Stable Colorectal Cancer, Pancreatic Cancer, or MSI High Colorectal Cancer.

The interventions involved in this study are:

* Nivolumab
* Ipilimumab
* Radiation Therapy

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved nivolumab for this specific disease but it has been approved for other uses.

The FDA (the U.S. Food and Drug Administration) has not approved ipilimumab for this specific disease but it has been approved for other uses.

Researchers hope to study the effects of the combination of Nivolumab and Ipilimumab. Many cancers use specific pathways (such as PD-1/PD-L1 and CTLA-4) to evade the body's immune system. Nivolumab and ipilimumab work by blocking the PD-1/PD-L1 and CTLA-4 pathways and thus releasing the brakes on the immune system so it can stop or slow cancer.

Ipilimumab and Nivolumab are both antibodies. An antibody is a cell that attaches to other cells to fight off infection. The antibodies in ipilimumab work by not allowing cancer cell growth. The antibodies in nivolumab work by causing programmed cell death of the cancer cells. Radiation therapy is believed to increase the likelihood of response of immunotherapy (the prevention/treatment of a disease through an immune response).

In this research study, the investigators are studying the combination of nivolumab, ipilimumab and radiation therapy on participants with microsatellite stable colorectal cancer, pancreatic cancer, or MSI high colorectal cancer. The combination of these study drugs have been tested and optimized for safety and is currently being tested in multiple disease types. The study drugs have not been tested and optimized in combination with radiation therapy. The investigators believe that through the combination of the study drugs and radiation therapy the body may produce an immune response to stop the cancer cells from growing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed adenocarcinoma of colorectal or pancreatic origin
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined in Table 1, all screening labs should be performed within 14 days of protocol registration.

Table 1 Adequate Organ Function Laboratory Values

System Laboratory Value

* Hematological

  * Absolute neutrophil count (ANC) ≥1500 /mcL
  * White blood count (WBC) ≥2000 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL
* Renal

  * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN (upper limit of normal) (subjects with Gilbert Syndrome can have a total bilirubin <3 mg/dL
  * aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and Alanine Aminotransferase ALT (SGPT) ≤ 3 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT)
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy
  * as long as PT or PTT is within therapeutic range of intended use of anticoagulants

    ≤1.5 X ULN unless subject is receiving anticoagulant therapy
  * as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine clearance should be calculated per institutional standard.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG)
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women who are not of childbearing potential, ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Ability to understand and the willingness to sign a written informed consent document.
* Stable dose of dexamethasone 2 mg or less for 7 days prior to initiation of treatment
* One previously unirradiated lesion amenable to radiotherapy 8 Gy x 3 and can meet dose constraints, and another unirradiated measurable lesion > 1 cm in size outside the radiation field that can be used as measurable disease
* Colorectal patients must have documentation of microsatellite status. Immunohistochemistry (IHC) is acceptable.
* Colorectal patients must have received prior Fluorouracil (5FU), Irinotecan and Oxaliplatin (any combination) or have a contraindication to receiving these agents.
* Pancreas patients must have progressed on at least 1 prior line of chemotherapy

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Participants who are receiving any other investigational agents.
* Patients are excluded if they have an active, known or suspected autoimmune disease other than those listed below. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Colorectal patients are excluded if they have had prior systemic treatment with an anti-CTLA4, anti-PD1 (Programmed cell death protein 1) or PDL1 (Programmed death-ligand 1) antibody. Pancreatic patients are excluded if they have previously received anti-CTLA-4 therapy. Prior PD-1 or PDL1 therapy will be permitted for pancreas patients
* Has a known history of active TB (Bacillus Tuberculosis)
* Patients are excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients are excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months for woman and 7 months for men, after the last dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled brain metastases. Patients treated with radiation > 4 weeks prior with follow up imaging showing control are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 2 years
  The percentage of participants with disease control following treatment with nivolumab/ipilimumab/radiation. Disease control is defined as the percentage of participants who have achieved complete response (CR), partial response (PR), or stable disease (SD) as defined by Response Evaluation Criteria In Solid Tumors (RECIST). Tumors may be evaluated for response with X-ray, computerized tomography (CT) scan, Magnetic resonance imaging (MRI), FDG (fluorodeoxyglucose) positron emission tomography (PET) scan, PET-CT, or cytology/histology.

SECONDARY OUTCOMES:
Median Progression free Survival | 2 years
  Progression-Free Survival (PFS) is defined as the time from the first treatment date to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Median Overall Survival | 2 years
  Overall Survival (OS) is defined as the time from the first treatment date to death due to any cause, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Koenig, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh AR, Szabolcs A, Allen JN, Clark JW, Wo JY, Raabe M, Thel H, Hoyos D, Mehta A, Arshad S, Lieb DJ, Drapek LC, Blaszkowsky LS, Giantonio BJ, Weekes CD, Zhu AX, Goyal L, Nipp RD, Dubois JS, Van Seventer EE, Foreman BE, Matlack LE, Ly L, Meurer JA, Hacohen N, Ryan DP, Yeap BY, Corcoran RB, Greenbaum BD, Ting DT, Hong TS. Radiation therapy enhances immunotherapy response in microsatellite stable colorectal and pancreatic adenocarcinoma in a phase II trial. Nat Cancer. 2021 Nov;2(11):1124-1135. doi: 10.1038/s43018-021-00269-7. Epub 2021 Nov 18. PMID 35122060